CLINICAL TRIAL: NCT01446263
Title: A Randomized Comparison of RADIAL Versus Femoral Access for Coronary Artery Bypass Graft Angiography and Intervention (RADIAL-CABG) Trial
Brief Title: RADIAL Versus Femoral Access for Coronary Artery Bypass Graft Angiography and Intervention (RADIAL-CABG) Trial
Acronym: RADIAL-CABG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Director, Cardiac Catheterization Laboratories, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: #11-063
Record Dates: First submitted 2011-09-29; First posted 2011-10-05 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Vascular Access Complication
Keywords: Radial access; Femoral access; Coronary angiography; Coronary artery bypass graft
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radial access (Active Comparator)
  Interventions: Procedure: Radial access versus femoral access for coronary angiography and intervention
- Femoral access (Active Comparator)
  Interventions: Procedure: Radial access versus femoral access for coronary angiography and intervention

INTERVENTIONS:
Procedure: Radial access versus femoral access for coronary angiography and intervention — Radial access or femoral access for coronary angiography and intervention in patients with prior coronary artery bypass grafts

SUMMARY:
Increased use of radial access for cardiac catheterization is being advocated because studies have showed lower arterial access related complication rates and higher patient satisfaction as compared to femoral access. However, little is known on patients with prior coronary artery bypass graft (CABG). The RADIAL CABG Trial is a randomized-controlled trial proposed to test the hypothesis that bypass graft angiography and intervention via radial access provides lower vascular complication rates, similar contrast and equipment utilization and higher patient satisfaction when compared with transfemoral approach.

DETAILED DESCRIPTION:
This is a phase III, single-center, prospective, randomized trial that will compare resource utilization, clinical outcomes and patient satisfaction between radial and femoral access for patients with prior coronary artery bypass graft (CABG)surgery undergoing coronary and graft angiography and intervention. During clinically-indicated coronary angiography of patients with prior CABG, the amount resources used, radiation exposure to patients and operators, occurence of complications and patients satisfaction will be compared between the two treatment arms to determine whether compared to femoral approach radial access will result in:

1. similar contrast utilization (primary endpoint)
2. similar procedure time (secondary endpoint)
3. similar fluoroscopy time (secondary endpoint)
4. similar radiation exposure of the patient - measured as DAP [dose area product] and AK [air kerma] (secondary endpoint)
5. similar radiation exposure of the operators using portable radiation dose measuring devices (secondary endpoint)
6. similar number and types of catheters and guidewires used (secondary endpoint)
7. reduction in vascular access complications (secondary endpoint)
8. reduction in overall complications (vascular access complications,injury, bleeding, death, emergency coronary bypass surgery, stroke, acute myocardial infarction) (secondary endpoint)
9. higher patient satisfaction as measured by standardized survey 24-hours after the procedure (secondary endpoint)

ELIGIBILITY:
Inclusion Criteria:

* Age >18-years
* Prior coronary artery bypass graft surgery
* Referred for clinically-indicated coronary and graft angiography and/or intervention
* Able to provide informed consent

Exclusion Criteria:

* Known pathologic Allen's test
* Known difficulty that limits vascular access at the femoral or radial arteries
* Age > 90

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Amount of contrast used | 24 hours

SECONDARY OUTCOMES:
Total procedure time | 24 hours
Fluoroscopy time | 24 hours
Radiation exposure of the patients measured as DAP [dose area product] and AK [air kerma] | 24 hours
Radiation exposure of the operators as measured as AK using portable radiation dose measuring devices | 24 hours
Performance of ascending aortic angiography to identify patent bypass grafts | 24 hours
Number of catheters and wires used | 24 hours
Vascular access complications (hematoma, aneurysm,pseudo-aneurysm, arterio-venous fistula formation, dissection, limb ischemia, bleeding) | 24 hours
Overall Complications (vascular access complications, injury, bleeding, death, emergency coronary bypass surgery, stroke, acute myocardial infarction) | 24 hours
Patient satisfaction, as measured by questionnaire administered 24 hours after the procedure | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil s Brilakis, MD, PhD, Principal Investigator — North Texas Veterans Healthcare System
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

REFERENCES:
- [Result] Michael TT, Alomar M, Papayannis A, Mogabgab O, Patel VG, Rangan BV, Luna M, Hastings JL, Grodin J, Abdullah S, Banerjee S, Brilakis ES. A randomized comparison of the transradial and transfemoral approaches for coronary artery bypass graft angiography and intervention: the RADIAL-CABG Trial (RADIAL Versus Femoral Access for Coronary Artery Bypass Graft Angiography and Intervention). JACC Cardiovasc Interv. 2013 Nov;6(11):1138-44. doi: 10.1016/j.jcin.2013.08.004. Epub 2013 Oct 16. PMID 24139930